CLINICAL TRIAL: NCT04914871
Title: Readiness for Basic Life Support in Schools: Randomized Controlled Trial
Brief Title: Readiness for Basic Life Support in Schools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 46377995
Record Dates: First submitted 2021-04-30; First posted 2021-06-07 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Health Education; First Aid; Cardiopulmonary Resuscitation
Keywords: Basic Life Support; Student; Teaching; Nursing; Readiness
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: According to the stated objectives, this study has a quantitative approach, Randomized Controlled Clinical Trial (RCT), with an experimental and control group and pre- and post-test measures; to explore the response of children to the intervention UN Lifeguard Kids in the Tunja version and approximation can be made its effectiveness.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research will be conducted using the double-blinded model since the children, parents, and research assistants who will carry out the pre- and post-test measurements, will not know the assignment of the groups, control, and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental protocol UN Lifeguard Kids in the Tunja version (Experimental): Group to which the experimental protocol will be offered.
  Interventions: Behavioral: Protocol UN Lifeguard Kids in the Tunja version
- Educational session, accident prevention and wound management. (Placebo Comparator): The control group will be offered the Educational session.
  Interventions: Behavioral: Educational session accident prevention and wound management

INTERVENTIONS:
Behavioral: Protocol UN Lifeguard Kids in the Tunja version — The experimental protocol UN Lifeguard Kids in the Tunja version done by the researcher following the guidelines of International organizations such as the American Heart association and European Resuscitation Council.
  The intervention consists of 3 sessions of 60 minutes of theoretical and practical exercises on BLS, developed within the usual class schedule.
  Arms: The experimental protocol UN Lifeguard Kids in the Tunja version
Behavioral: Educational session accident prevention and wound management — It will be provided to the control group
  Arms: Educational session, accident prevention and wound management.

SUMMARY:
This research is a response to problems with Cardiovascular Disease in Colombia, where circulatory system diseases are the first cause of mortality in the adult population, making them a critical issue for the country. It is known that around 70% of cardiac arrests occur outside health institutions, generally at home or on public roads.

To reduce these high mortality rates, international recommendations were issued to establish strategies to train the general population in cardiopulmonary resuscitation, especially school-age children. This constitutes a key stage for initiating learning. This condition significantly favors learning and preserving the acquired knowledge for the rest of their life.

Based on the reasons above, this pilot project seeks to be the first approach at the national level to train second-grade elementary school children in Basic Life Support. This training will describing the step by step experiences of the participants, focusing on: project viability related to recruitment and follow-up, acceptability, the experience of participation from the educational community, and the effects of implementing the intervention on the knowledge and skills in the child population. A virtual protocol will be implemented (adapted to the current situation generated by the Coronavirus pandemic), and will be developed through didactic methodologies in three 60-minute educational sessions, during regular class hours.

DETAILED DESCRIPTION:
1. Research question What are the viability, acceptability, and potential effects of implementing the UN Lifeguard Kids in the Tunja version intervention in two schools in the city of Tunja in 2021?
2. General objective:

   To describe the viability, acceptability, participation experience, and potential effects of implementing the UN Lifeguard Kids in the Tunja version intervention, in two schools in the city of Tunja in 2021.
3. Specific objectives To carry out the characterization of the child population under study. To describe the viability of the UN Lifeguard Kids in the Tunja version intervention in terms of recruitment and follow through.

   To describe the acceptability of the UN Lifeguard Kids in the Tunja version intervention for the child population that receives it.

   To describe the experience of participating in the UN Lifeguard Kids in the Tunja version intervention for the academic community.

   To describe the effects of the UN Lifeguard Kids in the Tunja version intervention on theoretical knowledge and practical skills in the child population that receives it.
4. A sample population of 70 children was determined as appropriate for the study. Two second-graded classes were selected to fulfill this requirement. Children were assigned to a control or test group using simple random sampling. Finally, five additional children were added to reduce sample attrition.
5. Biases control

   * Selection bias: It will be controlled in this study by strictly complying with the inclusion and exclusion criteria. Likewise, by applying the random blocks methodology for the allocation of the intervention and control group, guaranteeing an equitable distribution of children. Another measure is the application of the double-blind method so that neither the participants nor the research assistants responsible for measuring response variables, know which group they belong to or which intervention they received.
   * Detection biases: It will be controlled by including five nursing professionals who are not part of the study to carry out the measurements.
   * Attrition biases: There are two steps to control attrition. Firts, children will be motivated in each session through playful methodologies and novel didactic material, encouraging continued participation. Second, sessions will be within the usual class schedule to prevent abandonment.
   * Notification bias: It will be controlled through an ethical commitment by the researcher when publishing the complete results of the interventions. Additionally, these results will be publically available through the clinicaltrial.org portal.
   * Confusion biases: it will be controlled by randomization; distributing the known and unknown confounding variables equally between the groups and therefore, avoiding possible biases in the analysis. Subsequently, a comparison of the confounding variables will be made between the experimental and control groups before analyzing the response variables to identify the equivalence of the groups.
6. Statistical analysis: Descriptive statistics will be used for the analyses of the qualitative variables, through the distribution of frequencies and proportions. For continuous quantitative variables, descriptive statistics will be used with measures of central tendency (i.e. average and SD), dispersion, and 95% confidence intervals. For the intra- and inter-group comparisons of the continuous quantitative response variables, adjustment tests will be performed using the Kolgomorov Smirnov Gaussian model. If the adjustment is satisfactory, the comparisons will be made with paired Student's T-tests for intragroup and unpaired Student's T-tests for the intergroup analyses. Otherwise, Wilcoxon and Man Whitney U signed-rank tests will be performed, respectively.

ELIGIBILITY:
Inclusion criteria:

* Seven and eight-year-old.
* Children who are in the second grade of elementary school in two schools in the city of Tunja.
* Children's families with an available computer tablet or mobile device and internet connection will be considered for the study.
* Children who have a caregiver 18 years of age or older to accompany them during the intervention.
* Children with adequate learning skills (This data will be obtained from the report of the course teacher)

Exclusion criteria:

* Children who have received a scientific intervention on CPR.
* Children who participate in a rescue force (i.e., police, civil defense, brigade members).
* Children with a diagnosis of physical or mental disability (autism spectrum disorder, trisomy 21, Asperger syndrome, Tourette syndrome, attention deficit hyperactivity disorder (ADHD), severe visual, hearing, or motor problems, and/or similar disabilities).

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Viability | 8 weeks
  This variable is defined as the proportion of eligible participants who agree to participate in the study.
  Selection and monitoring form: In the first place, the form is filled out to discern if the children meet the inclusion criteria, then the consent form is signed, and finally the children agree to participate in the study.
  Then, the children who enter training sessions complete a form, in order to measure the percentage of children who attended all the sessions and to compare it with the children who were initially recruited.
Acceptability | 8 weeks
  Defined as the degree to which the participants were comfortable with their experience with the nursing intervention "UN Salvavidas Kids Tunja version".
  Participant's satisfaction questionnaire with the intervention: This approach has two parts, the first one involves three open questions and the second 6 with closed answers using dichotomous nominal variables.

SECONDARY OUTCOMES:
knowledge in Basic Life Support. | 8 weeks
  Defined as the initial measures to recognize, act and ask for help in an emergency. Questionnaire (it will be designed for researchers): evaluation of theoretical knowledge in basic Life support before and after intervention (8 weeks).
  It consists of 7 open questions with answers that are evaluated according to criteria (correct/incorrect response or fulfil/fails) that clarify which answers are eligible for scoring.
Skills in Basic Life Support. | 8 weeks
  Defined as the initial measures to recognize, act and ask for help in an emergency situation. Checklist (it will be designed for researchers): practical knowledge assessment in basic life support before and after intervention (8 weeks): It is done in a simulated situation in which children must apply the knowledge acquired during the training.
  It consists of 6 questions, each one has a statement and an administration condition that must be followed as described and a scoring criterion that clarifies what behavior is acceptable to receive a score(correct/incorrect action for fulfil/fails).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Patricia Carreño Moreno, RN, MSc, PhD, Study Director — Universidad Nacional de Colombia

IPD SHARING:
Plan to Share IPD: Yes
After data analysis, using the results obtained in this study, and the generation of the final report, the database will be shared shared with the public.
Supporting Information: SAP, ICF, CSR
Time Frame: five years.
Access Criteria: Access Criteria:
  Health workers and researchers. Nursing students. Health science students. Research teachers. Students in education. Applications will be received by email from the researcher lucanor@unal.edu.co, where an analysis will be carried out to share the information on the intervention.

REFERENCES:
- [Background] Bottiger BW, Van Aken H. Training children in cardiopulmonary resuscitation worldwide. Lancet. 2015 Jun 13;385(9985):2353. doi: 10.1016/S0140-6736(15)61099-6. No abstract available. PMID 26088639
- [Background] Yasunaga H, Horiguchi H, Tanabe S, Akahane M, Ogawa T, Koike S, Imamura T. Collaborative effects of bystander-initiated cardiopulmonary resuscitation and prehospital advanced cardiac life support by physicians on survival of out-of-hospital cardiac arrest: a nationwide population-based observational study. Crit Care. 2010;14(6):R199. doi: 10.1186/cc9319. Epub 2010 Nov 4. PMID 21050434
- [Background] Semeraro F, Wingen S, Schroeder DC, Ecker H, Scapigliati A, Ristagno G, Cimpoesu D, Bottiger BW. KIDS SAVE LIVES-Three years of implementation in Europe. Resuscitation. 2018 Oct;131:e9-e11. doi: 10.1016/j.resuscitation.2018.08.008. Epub 2018 Aug 8. No abstract available. PMID 30098386
- [Background] Oving I, Masterson S, Tjelmeland IBM, Jonsson M, Semeraro F, Ringh M, Truhlar A, Cimpoesu D, Folke F, Beesems SG, Koster RW, Tan HL, Blom MT; ESCAPE-NET Investigators. First-response treatment after out-of-hospital cardiac arrest: a survey of current practices across 29 countries in Europe. Scand J Trauma Resusc Emerg Med. 2019 Dec 16;27(1):112. doi: 10.1186/s13049-019-0689-0. PMID 31842928